CLINICAL TRIAL: NCT05945810
Title: Evaluation of TLL-018 Extended Release Formulation (ER, 50 mg QD) and TLL-018 Immediate-release Formulation (IR, 20 mg BID) for Human Bioequivalence Testing in Single Dose and Steady State in Healthy Chinese Subjects
Brief Title: Evaluation of TLL-018 Extended and Immediate Release Formulation for Bioequivalence Testing in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Highlightll Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TLL-018-103
Record Dates: First submitted 2023-07-05; First posted 2023-07-14 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis
Keywords: Bioequivalence; Extended Release tablet
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Eligible subjects screened will be randomly assigned to sequence A and sequence B in a 1:1 ratio. In cycle 1, subjects in sequence A receive a 50-mg single dose of TLL-018 extended-release tablet on day 1, and once daily for 5 consecutive days from day 3 onwards. After a 3-day washout period, subjects enter the cycle 2 at day 11 when they receive a 20-mg single dose of TLL-018 immediate-release tablet on the morning and another dose 12 hours later at night. From day 13 onward, they continue to receive 20 mg TLL-018 immediate-release tablets twice daily for 5 consecutive days. The subjects will be hospitalized for observation for 3 days after the end of medication.
  Subjects randomly assigned to sequence B received 20 mg of TLL-018 immediate-release tablets in cycle 1 and 50 mg extended-release tablet in cycle 2. The medication pattern was consistent with that of the subjects in sequence A. All the subjects took medicine after meal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sequence A (Experimental): In cycle 1, subjects in sequence A receive a 50-mg single dose of TLL-018 extended-release tablet on day 1, and once daily for 5 consecutive days from day 3 onwards. After a 3-day washout period, subjects enter the cycle 2 at day 11 when they receive a 20-mg single dose of TLL-018 immediate-release tablet on the morning and another dose 12 hours later at night. From day 13 onward, they continue to receive 20 mg TLL-018 immediate-release tablets twice daily for 5 consecutive days.
  Interventions: Drug: TLL-018 extended-release tablet; Drug: TLL-018 immediate-release tablet
- sequence B (Experimental): In cycle 1, subjects in sequence B receive a 20-mg single dose of TLL-018 immediate-release tablet on the morning on day 1 and another dose 12 hours later at night. From day 3 onward, they continue to receive 20-mg TLL-018 immediate-release tablets twice daily for 5 consecutive days. After 3 days of washout, subjects receive a 50-mg single dose of TLL-018 extended-release tablet on day 11 In cycle 2, and once daily for 5 consecutive days from day 13 onwards.
  Interventions: Drug: TLL-018 extended-release tablet; Drug: TLL-018 immediate-release tablet

INTERVENTIONS:
Drug: TLL-018 extended-release tablet — 50mg TLL-018 extended-release tablet QD
  Other Names: extended-release tablet
Drug: TLL-018 immediate-release tablet — 20mg TLL-018 immediate-release tablet BID
  Other Names: immediate-release tablet

SUMMARY:
The goal of this two-sequence, two-cycle, single and multiple-dose Phase I clinical trial is To evaluate the human bioequivalence of the test preparation and the reference preparation in 28 healthy chinese subjects at a single center.

DETAILED DESCRIPTION:
The goal of this two-sequence, two-cycle, single and multiple-dose Phase I clinical trial is To evaluate the human bioequivalence of the test preparation and the reference preparation in 28 healthy chinese subjects at a single center.

The main questions it aims to answer are:

* Sectionalization - subjects are divided into two sequences (A/B) equally of 14 subjects each
* Phases - The study is divided into 4 phases, screening, cycle 1, cycle 2 and follow-up observation period. The screening period is from D-7 to D-1, with subjects admitted to the phase I clinical trial ward at D-1. D1 starts the first cycle of the trail until D7 ends; After a 3-day washout period, D11 begins the second cycle of administration until D17 ended. D18~D20 are the follow-up observation period. The total study duration is 27 days.
* Medication - All subjects were administered after meal.

Participants in sequence A will receive oral administration of 50 mg TLL-018 extended-release tablet once on day 1 for the first cycle, and then continue to receive the same dosage once daily for 5 consecutive days from day 3. After a 3-day washout period, they will enter the second cycle and will receive one oral dose of 20 mg TLL-018 immediate-release tablet in the morning of day 11, followed by a second dose of 20 at night 12 hours later, then continued to receive 20 mg TLL-018 twice daily for 5 consecutive days from day 13. Hospital observation for 3 days after taking the medication..

Participants in sequence B will receive 20 mg TLL-018 immediate-release tablet in the first cycle and 50 mg TLL-018 extended-release tablet in the second cycle, with the same medication pattern as those in sequence A.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects can fully understand the purpose, method and possible adverse event of the study and are willing to participate and sign informed consent form prior to any study procedure;
2. 18-45 years (including 18 and 45 years);
3. weigh: Male ≥50.0 kg, female ≥ 45.0kg, BMI between 19.0 and 26.0 kg/m2 (including boundary value);
4. Without chronic or serious diseases history in cardiovascular, liver, kidney, blood and lymphatic, endocrine, immune, spiritual, menstrual and gastrointestinal systems, without dysphagia or any other effects on drug absorption history, no family history of genetic disease, and generally in good health;
5. Vital signs examination (including boundary value) : systolic blood pressure 90~139mmHg, diastolic blood pressure 60-89 mmHg, pulse 55-100 beats/min, body temperature (ear temperature) 36.0~37.4℃. Physical examination, clinical laboratory examination, 12-lead electrocardiogram, anterolateral chest radiograph, Abdominal B-ultrasonography results all show no abnormality or no clinical significance;
6. Female subjects are non-pregnant or non-lactating, and subjects and their partners are voluntary use of contraception deemed effective by the investigator for at least 4 weeks after the last investigational drug ;
7. The subject is able to communicate well with the investigator and understand and comply with all aspects of the study.

Exclusion Criteria:

1. People with a history of allergies, including but not limited to research drugs, foods or other substances;
2. Any history of surgery, trauma that may affect the safety of the study or the in vivo course of the drug, or Patients scheduled to undergo surgery during the study period;
3. Active or latent or inadequately treated mycobacterium tuberculosis infection in the 3 months prior to screening;
4. Patients with clinically significant symptoms of infection within 30 days prior to screening or acute illness prior to the use of the investigational drug.
5. Subjects with a history of herpes zoster within 1 year prior to screening; Subjects with a history of recurrent (unlimited) herpes zoster or disseminated herpes simplex or herpes zoster (even if only once);
6. Those who received vaccination within 30 days prior to screening or planned to receive vaccination during the study period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Single Dose: AUC0-t | Screening up to Day 17
  Area under the blood concentration-time curve from time 0 to the last measurable time t after dosing
Single Dose: AUC0-∞ | Screening up to Day 17
  Area under the blood concentration-time curve from time 0 to infinity after dosing
stable state: AUC0-24 | Screening up to Day 17
  Area under the blood concentration-time curve from time 0 to 24 hours after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No